CLINICAL TRIAL: NCT01513200
Title: A Two Part Study to Assess the Pharmacodynamic Effects of Unfractionated Heparin (UFH) in Healthy Volunteers and the Effects of Bendavia™ and Unfractionated Heparin When Administered Concurrently
Brief Title: Study to Assess the Pharmacodynamic Effects of Unfractionated Heparin (UFH) in Healthy Volunteers With and Without Bendavia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SPIRI-155
Record Dates: First submitted 2012-01-06; First posted 2012-01-20 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Heparin; arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- UFH + Placebo (Placebo Comparator): UFH (60U/kg bolus followed by 12U/kg/hr for approx.11 hours) with saline (placebo) administered as infusion for the last 4 hours of UFH
  Interventions: Drug: Unfractionated heparin (UFH); Drug: Saline (0.9%, sterile, for infusion)
- UFH + Bendavia (Experimental): UFH (60U/kg bolus followed by 12U/kg/hr for approx.11 hours) with Bendavia (0.25mg/kg/hr) administered as infusion for the last 4 hours of UFH
  Interventions: Drug: Unfractionated heparin (UFH); Drug: Bendavia

INTERVENTIONS:
Drug: Unfractionated heparin (UFH) — UFH solution for infusion Initially 60U/kg bolus followed by intravenous infusion (12U/kg/hr) for approximately 11 hours
Drug: Bendavia — Bendavia for infusion Constant intravenous infusion (Bendavia 0.25mg/kg/hr) for 4 hours
  Arms: UFH + Bendavia
Drug: Saline (0.9%, sterile, for infusion) — Saline (placebo) Constant IV infusion for 4 hours
  Arms: UFH + Placebo

SUMMARY:
This will be a phase 1 randomized, double-blind crossover trial enrolling approximately 12 healthy volunteers to assess whether intravenous (IV) UFH and IV Bendavia administered together have any significant impact on the pharmacodynamic effects of UFH and the pharmacokinetics of Bendavia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females aged between 18 and 65 years of age with signed informed consent.
* Women who are not post-menopausal (without menstrual bleed for >24 months) or surgically sterile must have a negative serum pregnancy test at screening and within 24 hours of treatment with understanding (through informed consent process) to not become pregnant over the duration of the study and must agree to employ an effective form of birth control for the duration of the study [Acceptable forms of birth control are: double-barrier contraceptives (condom, diaphragm with spermicide) or intra-uterine device (IUD) 1 week prior to and at least 30 days post treatment even if hormonal contraceptives are used]

Exclusion Criteria:

* Serum sodium level below the lower limit of the site's clinical laboratory normal range at both study period qualification visits,
* Platelet value below the lower limit of normal range at screening or admission,
* aPTT value outside the normal range at screening or admission,
* Creatinine clearance calculated by the Cockcroft and Gault method calculated to be <90 mL/min for males and <80 mL/min for females,
* Any addition laboratory abnormalities determined as clinically significant by the Principal Investigator at laboratory screening,
* Clinically significant abnormalities on physical examination,
* Body Mass Index (BMI) of less than 18 kg/m2 or greater than 32 kg/m2,
* Any disease or condition that might compromise the cardiovascular, hematological, renal, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous, or gastrointestinal (including an ulcer) systems,
* History of seizures or history of epilepsy,
* History of serious (Principal Investigator judgment) mental illness,
* Receipt of investigational medicinal product within 30 days before planned date of unfractionated heparin and/or study drug administration,
* Positive serology for human immunodeficiency virus 1 or 2 (HIV1 or 2), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV),
* Fever greater than 37.5°C at the time of planned dosing,
* Suspicion of or recent history of alcohol or substance abuse,
* Donated blood or blood products within the past 30 days,
* Women who are pregnant or breastfeeding,
* Employee or family member of the investigational site,
* Subjects who currently smoke cigarettes, cigars, pipes or chew tobacco products or who have used any tobacco products in the 30 days prior to screening,
* Subjects who are either unwilling to agree to refrain from using or found to be using:

  1. Alcohol, caffeine, xanthine-containing food or beverages, nicotine products and over-the-counter medications with the exception of Tylenol from 24 hours prior to dosing and throughout the confinement period
  2. Prescription medications from 14 days prior to and 7 days post treatment (excluding hormonal contraceptives)
  3. Hormonal contraceptives without concomitant use of double-barrier contraceptives (condom, diaphragm with spermicide) for a period of 7 days prior to and 30 days post treatment
* Subjects taking aspirin or any other non-steroidal anti-inflammatory agent, either prescription or over-the-counter, within 10 days of treatment,
* Subjects known to have allergic or untoward effects when using unfractionated heparin,
* Subjects having previous exposure to Bendavia,
* Subjects who are expected to undergo any surgical procedure within 14 days of the completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Mean difference over 24 hours in aPTT (activated partial prothrombin time) in seconds when UFH is administered with and without Bendavia | Pre-UFH to 24 hours post-study drug administration
  Difference in group (with/without Bendavia) means of aPPT values will be assessed for statistical significance (Analysis of Variance; ANOVA) at the following time points:
  Pre-UFH, Pre-Study-Drug infusion start and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours Post-Study-Drug infusion start.

SECONDARY OUTCOMES:
Mean difference over 12 hours of anti-factor Xa (IU/mL) when UFH is administered with and without Bendavia | Pre-UFH to 12 hours post-study drug administration
  Difference in group (with/without Bendavia) means of aPPT values will be assessed for statistical significance (ANOVA) at the following time points:
  Pre-UFH, Pre-Study-Drug infusion start and 4, 8 and 12 hours Post-Study-Drug infusion start.
Mean difference in Bendavia Area Under the Curve(0-infinity) (AUC) when Bendavia is administered with and without UFH (historical data will be used to provide bendavia without UFH) | 48 hours post-study-drug administration
Difference in number of adverse events when UFH is administered with and without Bendavia | Pre-dose through Day 10
  Adverse events will be described by treatment group (UFH with and without Bendavia). No statistical analysis of the difference between AEs will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Lasseter, MD, Principal Investigator — Clinical Pharmacology of Miami; Richard Straube, MD, Study Director — Stealth Peptides
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States